CLINICAL TRIAL: NCT06612450
Title: Turbinate Volume Reduction Under Local Anesthesia: Randomized Clinical Trial; Our Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ibrahim M. Gehad, Dr. Ibrahim Gehad, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU200-289
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Nasal Obstruction; Turbinate Surgery
Keywords: Turbinate Hypertrophy; Coblation; Radiofrequency; Nasal obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: only one surgeon did the surgeries, other two assessors didnt know which intervention was done, the patient didn't know which group did they belong to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coblation (Active Comparator): patients will undergo turbinoplasty using coblation wand
  Interventions: Device: turbinate surgery
- RaVoR (Active Comparator): patients will undergo turbinate reduction using ravor radiofrequency
  Interventions: Device: turbinate surgery

INTERVENTIONS:
Device: turbinate surgery — Turbinoplasty to decrease the turbinate size in cases with turbinate hypertrophy with mainly soft tissue component without sacrificing the mucosal function

SUMMARY:
The purpose of this trial is to know which method is better in delivering radiofrequency waves for hypertrophied turbinates: coblation or RavoR technique? Researchers will compare both techniques in randomized blinded manner patients will have subjective outcomes like NOSE score, pain Objective outcomes like Turbinate size over long term clinical follow up visits for 1 year

ELIGIBILITY:
Inclusion Criteria:

All patients with the following criteria were eligible for inclusion:

1. Age group: 18-60 years old.
2. Patients complaining of chronic nasal obstruction because of bilateral (HIT) diagnosed by our former protocol refractory to medical treatment for at least three months.
3. Evident (HIT) on the CT nose and paranasal sinuses with mainly soft tissue component hypertrophy with or without minimal septal deviation without any other cause for the obstruction.
4. Patients who are unfit for general anesthesia

Exclusion Criteria:

* All Patients with:

Marked septal deviation or Concha Bullosa, Nasal polyps, Sinonasal Tumors, Any previous nasal surgeries or radiotherapy, Chronic sinusitis or Cystic Fibrosis, Pregnancy, Patients with severe bleeding tendency, coagulopathy disorder, and Patients who refuse participation in this study were excluded from our study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
NOSE score | 1 year
  nasal obstruction symptom score for subjective analysis of patient symptom before and after intervention
Pain VAS score | 1-3 months postoperative
  patient score on a scale from 0 to 10 where 0 is no pain and 10 is most severe pain
Turbinate Size grading | 1 year postoperative
  endoscopic grading of turbinate size before and after intervention from 0-4 where 1 is 25% of nasal cavity

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El-Sheikh Universitty, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be shared with results
Supporting Information: Study Protocol, SAP
Time Frame: when results are finalized will be available for 6 months